CLINICAL TRIAL: NCT01898871
Title: Using Indigenous Foods to Reduce Malnutrition in Children
Brief Title: Effectiveness of Nutritional Products to Treat Moderate Acute Malnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Food and Nutrition Research, Yaounde (Other Government)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Medoua Nama Gabriel, Deputy Head of Centre, Centre for Food and Nutrition Research, Yaounde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMR6010
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Wasting; Moderate Acute Malnutrition
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ready to Use Suplementary Food (RUSF) (Experimental): A daily ration of 40 kcal/kg of body weight during 56 days
  Interventions: Dietary Supplement: A daily ration of 40 kcal/kg of body weight during 56 days
- Corn Soya Blend (CSB+) (Active Comparator): A daily ration of 40 kcal/kg of body weight during 56 days
  Interventions: Dietary Supplement: A daily ration of 40 kcal/kg of body weight during 56 days

INTERVENTIONS:
Dietary Supplement: A daily ration of 40 kcal/kg of body weight during 56 days — On enrollment, children were examined by a pediatrician to assess their health status and they were de-wormed with one tablet of Mebendazole 500 mg.

SUMMARY:
The purpose of this study is to determine whether an improved corn-soya blend (CSB+) and a new formulated ready-to-use supplementary food (RUSF) are effective in the treatment of moderate acute malnutrition in children.

DETAILED DESCRIPTION:
Assuming the availability of some food in the household, the caregivers were instructed on how best to use the food they have and the quantity of supplementary food distributed was calculated to provide about 50% of child energy requirement.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-59 month
* Weight-for-height between -3 and -2 z-scores without edema
* Good appetite
* Stable clinical conditions

Exclusion Criteria:

* Weight-for-Height Z-score < -3
* Presence of bilateral pitting edema
* Unstable clinical conditions
* Not showing appetite

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Recovery rate of the children receiving CSB+ or RUSF | 56 days
  Children with Weight-for-Height Z-score > -2

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Medoua Nama, Ph.D., Principal Investigator — Centre for Food and Nutrition Research, IMPM
Locations (2):
- Cameroon (2):
  - Evodoula Health District, Évodoula
  - Biyem Assi District Centre, Yaoundé